CLINICAL TRIAL: NCT03753633
Title: Efficiency of Speech Therapy in Resistant Hypertensive Patients With Mild Obstructive Sleep Apnea Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Alessandra Bastos de Sousa, Master student, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 62061716.1.0000.5257
Record Dates: First submitted 2017-01-26; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Sleep Apnea, Obstructive; Hypertension Secondary
Keywords: speech therapy; sleep apnea; resistant hypertension; quality of life; quality of sleep
MeSH Terms: conditions — Sleep Apnea, Obstructive; Communication Disorders; Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Speech therapy Group (Experimental): 25 patients will be treated with speech therapy, once a week, during 40 minutes for 12 weeks. Oropharyngeal exercises will be performed under the supervision of a speech therapist. Patients will perform the oropharyngeal exercises at home every day.
  Interventions: Other: Speech therapy
- Control Group (Sham Comparator): 25 patients will perform inspiratory and expiratory exercises recruiting diaphragmatic muscle.
  Interventions: Other: Control

INTERVENTIONS:
Other: Speech therapy — Oropharyngeal exercises will be performed under the supervision of a speech therapist.
  Arms: Speech therapy Group
Other: Control — Inspiratory and expiratory exercises recruiting diaphragmatic muscles
  Arms: Control Group

SUMMARY:
The purpose of this study is to analyze the effect of speech therapy on quality of life, sleep quality, daytime sleepiness level and apnea-hypopnea index in patients with hypertensive patients with mild obstructive apnea syndrome.

DETAILED DESCRIPTION:
The database will include demographic characteristics, cardiovascular risk factors and and target-organ damages. Anthropometric measurements (height, weight, and abdominal and neck circumference) will be registered. Daytime sleepiness, quality of sleep and quality of life wiill be evaluated through the respective questionnaires: Epworth sleepiness scale, Pittsburgh Sleep Quality Index (PSQI) and SF-36. In order to evaluate the airway, the Mallampati grade will be used in addition to the adapted assessment protocol from Guimarães (2009). The differences between the final score and the baseline score will be calculated and adjusted by the baseline value found in each of the questionnaires applied. Finally, the analysis excluding the patients with suboptimal adherence to speech therapy treatment (less than 85%) compared to the control group will be redone. If there are benefits of treatment with speech therapy, it will also be offered to the control group after the end of the clinical trial. Statistical analysis will be done in the statistical package SPSS version 19.0 package (SPSS Inc. Chicago, Illinois, USA). Data obtained may be of benefit to future patients and will be used only for statistical purposes. The confidentiality of the information collected will be guaranteed, thus ensuring the privacy and confidentiality of the information. In addition, the data obtained will not be used for other purposes not foreseen in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients in follow-up in the Hypertension Program (ProHart) at Hospital Universitário Clementino Fraga Filho - UFRJ at least six months;
* Patient with Resistant Hypertension and Mild Obstructive Sleep Apnea detected by polysomnography;
* All participants that give written informed consent.

Exclusion Criteria:

* Age> 85 years;
* Cognitive deficit that prevents speech therapy;
* Severe clinical events in the last 6 months;
* Refusal of the patient to participate in the study;
* Pregnancy;
* Prior and regular use of CPAP;
* Clinical data suggestive of neurological disease with cognitive and / or motor sequelae, craniofacial malformation, severe upper airway obstruction, Neuromuscular disease, users of hypnotic drugs

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Epworth sleepiness scale | Five months
  Changes found in score after 12 weeks in control group and speech therapy group. The ESS measures EDS levels, assigning a score (from 0 to 3) according to the possibility of sleeping in each mentioned situation. A score from 0 to 6 is considered normal; from 7 to 9, limitrophe; 10 to 14, mild sleepiness; 15 to 20, moderate sleepiness; and above, severe sleepiness. Values ≥11 are generally associated with sleep disorders.
Changes in SF-36 | Five months
  Changes found in score after 12 weeks in control group and speech therapy group. The SF-36 consisting of 36 items grouped into eight domains: functional capacity, physical aspects, pain, general health status, vitality, social aspects, emotional aspects and mental health. It assesses both negative (illness or disease) and positive aspects (well-being), with a score from 0 to 100, with zero being the worst health condition and 100 being the best, with each dimension being analyzed separately.
Changes in Pittsburgh Sleep Quality Index (PSQI) | Five months
  Changes found in score after 12 weeks in control group and speech therapy group. O questionário de Pittsburgh permite avaliar o sono de forma qualitativa e quantitativa, de forma padronizada, ao determinar os "bons dormidores" e "maus dormidores". O questionário avalia parâmetros quantitativos, tais como a duração do sono, latência do sono e número de despertares; e parâmetros qualitativos, que são puramente subjetivos.

SECONDARY OUTCOMES:
Apnea-hypopnea index | Three months after Clinical evaluation initial
  The patients were submitted to polysomnography using BrainNet BNT Polipolygraph, supervised by a qualified professional. Electroencephalogram, electrooculogram, submental electromyogram, nasal airflow, oximetry, respiratory effort, electrocardiogram and anterior tibial electromyogram were realized. The exam was complemented with video monitoring. Patients who had less than 240 minutes of sleep in the night were excluded.The report was prepared by a qualified medical professional, Sleep Medicine specialist and with a practice certificate in the area, who was unaware of the patients; clinical data, according to the norms established in the American Academy of Sleep Medicine manual.
Qualitative assessment of Speech Therapy Assessment | Four months
  Changes in Orofacial Myofunctional after speech therapy in therapy group and after 12 weeks after the evaluation initial in control group. Data were collected from the oromiofunctional speech-language assessment protocol, with face evaluation (eyes, nostrils, lips, cheeks, jaw, tongue and palate) and functions (breath, chew and speech). The UAW physical status, evaluated through the modified Mallampati classification, checks according to the spatial relationship between the soft palate and the body of tongue with the pharynx posterior wall and the narrowing of veil and hypopharynx( class 1, the entire palatopharyngeal veil and uvula are visualized; class 2, uvula and palatopharyngeal veil arches partially visualized; class 3, uvula or palatopharyngeal veil not visualized; class 4, all soft palate not visualized). The anthropometric measurements: height and weight to calculate BMI, neck circumference(greater than 41 cm - women - and 43 cm - men) and waist circumference.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra B de Sousa, Principal Investigator — Universidade Federal do Rio de Janeiro; Mariana P Brendim, Master, Study Chair — Universidade Federal do Rio de Janeiro; Elizabeth S Muxfeldt, Study Director — Universidade Federal do Rio de Janeiro
Locations (1):
- Hospital Universitário Clementino Fraga Filho, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AASM - American Academy of Sleep Medicine, International Classification of Sleep Disorders: diagnostic and coding manual, 2nd ed. Westchester, Ill: American Academy of Sleep Medicine; 2005.
- [Background] Acelajado MC, Calhoun DA. Aldosteronism and resistant hypertension. Int J Hypertens. 2011 Jan 20;2011:837817. doi: 10.4061/2011/837817. PMID 21331160
- [Background] Barnes M, Houston D, Worsnop CJ, Neill AM, Mykytyn IJ, Kay A, Trinder J, Saunders NA, Douglas McEvoy R, Pierce RJ. A randomized controlled trial of continuous positive airway pressure in mild obstructive sleep apnea. Am J Respir Crit Care Med. 2002 Mar 15;165(6):773-80. doi: 10.1164/ajrccm.165.6.2003166. PMID 11897643
- [Background] Berger G, Berger R, Oksenberg A. Progression of snoring and obstructive sleep apnoea: the role of increasing weight and time. Eur Respir J. 2009 Feb;33(2):338-45. doi: 10.1183/09031936.00075408. Epub 2008 Nov 14. PMID 19010989
- [Background] Berry RB, Gamaldo CE, Harding SM et al. The AASM Manual for the Scoring of Sleep and Associated Events: Rules, Terminology and Technical Specifications, Version 2.2. www.aasmnet.org. Darien, Illinois: Am Acad Sleep Med, 2015.
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Dartora EG, Miozzo IC, de Barba ME, Barreto SS. Validation of the Brazilian Portuguese version of the Pittsburgh Sleep Quality Index. Sleep Med. 2011 Jan;12(1):70-5. doi: 10.1016/j.sleep.2010.04.020. Epub 2010 Dec 9. PMID 21145786
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Pedro VD, Menna Barreto SS, Johns MW. Portuguese-language version of the Epworth sleepiness scale: validation for use in Brazil. J Bras Pneumol. 2009 Sep;35(9):877-83. doi: 10.1590/s1806-37132009000900009. English, Portuguese. PMID 19820814
- [Background] Bittencourt LRA, Togeiro SMGP, Bagnato MC. Diagnóstico da síndrome da apnéia e hipopnéia obstrutiva do sono. In: Stamm A. ed. Rinologia; 2002. São Paulo: Komedi, 2002: 103-111. Disponível em:<http://www.moreirajr.com.br/revistas.asp?fase=r003&id_materia=1628>
- [Background] Bloch KV, Melo AN, Nogueira AR. [Prevalence of anti-hypertensive treatment adherence in patients with resistant hypertension and validation of three indirect methods for assessing treatment adherence]. Cad Saude Publica. 2008 Dec;24(12):2979-84. doi: 10.1590/s0102-311x2008001200030. Portuguese. PMID 19082292
- [Background] Brown LK. Mild obstructive sleep apnea syndrome should be treated. Pro. J Clin Sleep Med. 2007 Apr 15;3(3):259-62. No abstract available. PMID 17561591
- [Background] Burger RCP, Caixeta EC, Di Ninno CQMS. A relação entre apnéia do sono, ronco e respiração oral. Rev CEFAC 2004; 6(3):266-271. Disponível em: <http://cefac.br/revista/revista63/Artigo%206.pdf>.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Calhoun DA, Jones D, Textor S, Goff DC, Murphy TP, Toto RD, White A, Cushman WC, White W, Sica D, Ferdinand K, Giles TD, Falkner B, Carey RM. Resistant hypertension: diagnosis, evaluation, and treatment. A scientific statement from the American Heart Association Professional Education Committee of the Council for High Blood Pressure Research. Hypertension. 2008 Jun;51(6):1403-19. doi: 10.1161/HYPERTENSIONAHA.108.189141. Epub 2008 Apr 7. PMID 18391085
- [Background] Chung F, Abdullah HR, Liao P. STOP-Bang Questionnaire: A Practical Approach to Screen for Obstructive Sleep Apnea. Chest. 2016 Mar;149(3):631-8. doi: 10.1378/chest.15-0903. Epub 2016 Jan 12. PMID 26378880
- [Background] Ciconelli RM. et al. Tradução para o português e validação do questionário genérico de avaliação de qualidade de vida "medical outcome study 36-item shortform health survey (SF-36)". Tese (Doutorado em Reumatologia) - Universidade Federal de São Paulo, São Paulo; 1997. Disponível em: http://www.nutrociencia.com.br/upload_files/ artigos_download/qualidade.pdf.
- [Background] Cushman WC, Ford CE, Cutler JA, Margolis KL, Davis BR, Grimm RH, Black HR, Hamilton BP, Holland J, Nwachuku C, Papademetriou V, Probstfield J, Wright JT Jr, Alderman MH, Weiss RJ, Piller L, Bettencourt J, Walsh SM; ALLHAT Collaborative Research Group. Success and predictors of blood pressure control in diverse North American settings: the antihypertensive and lipid-lowering treatment to prevent heart attack trial (ALLHAT). J Clin Hypertens (Greenwich). 2002 Nov-Dec;4(6):393-404. doi: 10.1111/j.1524-6175.2002.02045.x. PMID 12461301
- [Background] Dantas RA, Sawada NO, Malerbo MB. [Research on quality of life: review of the scientific production of public universities from the state of Sao Paulo]. Rev Lat Am Enfermagem. 2003 Jul-Aug;11(4):532-8. doi: 10.1590/s0104-11692003000400017. Portuguese. PMID 14748173
- [Background] Daugherty SL, Powers JD, Magid DJ, Tavel HM, Masoudi FA, Margolis KL, O'Connor PJ, Selby JV, Ho PM. Incidence and prognosis of resistant hypertension in hypertensive patients. Circulation. 2012 Apr 3;125(13):1635-42. doi: 10.1161/CIRCULATIONAHA.111.068064. Epub 2012 Feb 29. PMID 22379110
- [Background] de Souza F, Muxfeldt ES, Salles GF. Prognostic factors in resistant hypertension: implications for cardiovascular risk stratification and therapeutic management. Expert Rev Cardiovasc Ther. 2012 Jun;10(6):735-45. doi: 10.1586/erc.12.58. PMID 22894630
- [Background] Dudenbostel T, Calhoun DA. Resistant hypertension, obstructive sleep apnoea and aldosterone. J Hum Hypertens. 2012 May;26(5):281-7. doi: 10.1038/jhh.2011.47. Epub 2011 Jun 9. PMID 21654850
- [Background] Epstein LJ, Kristo D, Strollo PJ Jr, Friedman N, Malhotra A, Patil SP, Ramar K, Rogers R, Schwab RJ, Weaver EM, Weinstein MD; Adult Obstructive Sleep Apnea Task Force of the American Academy of Sleep Medicine. Clinical guideline for the evaluation, management and long-term care of obstructive sleep apnea in adults. J Clin Sleep Med. 2009 Jun 15;5(3):263-76. PMID 19960649
- [Background] Finn L, Young T, Palta M, Fryback DG. Sleep-disordered breathing and self-reported general health status in the Wisconsin Sleep Cohort Study. Sleep. 1998 Nov 1;21(7):701-6. PMID 11286346
- [Background] Friedman M, Wilson MN, Pulver T, Pandya H, Joseph NJ, Lin HC, Chang HW. Screening for obstructive sleep apnea/hypopnea syndrome: subjective and objective factors. Otolaryngol Head Neck Surg. 2010 Apr;142(4):531-5. doi: 10.1016/j.otohns.2009.12.038. PMID 20304273
- [Background] Genta-Pereira DC, Pedrosa RP, Lorenzi-Filho G, Drager LF. Sleep disturbances and resistant hypertension: association or causality? Curr Hypertens Rep. 2014 Aug;16(8):459. doi: 10.1007/s11906-014-0459-3. PMID 24913922
- [Background] Giles TL, Lasserson TJ, Smith BJ, White J, Wright J, Cates CJ. Continuous positive airways pressure for obstructive sleep apnoea in adults. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD001106. doi: 10.1002/14651858.CD001106.pub2. PMID 16437429
- [Background] Guimarães K. Alterações no tecido mole de orofaringe em portadores da apnéia do sono obstrutiva. J Bras Fonoaudiol 1999; 1:69-75. Disponível em: <http://www.cefac.br/library/teses/48cf76d0f5fcc9cd822dc3a8bf181974.pdf>.
- [Background] Guimarães, KCC. Apnéia e Ronco: Tratamento Miofuncional Orofacial. São José dos Campos: Pulso; 2009.
- [Background] Hla KM, Young TB, Bidwell T, Palta M, Skatrud JB, Dempsey J. Sleep apnea and hypertension. A population-based study. Ann Intern Med. 1994 Mar 1;120(5):382-8. doi: 10.7326/0003-4819-120-5-199403010-00005. PMID 8304655
- [Background] Hu X, Fan J, Chen S, Yin Y, Zrenner B. The role of continuous positive airway pressure in blood pressure control for patients with obstructive sleep apnea and hypertension: a meta-analysis of randomized controlled trials. J Clin Hypertens (Greenwich). 2015 Mar;17(3):215-22. doi: 10.1111/jch.12472. Epub 2015 Jan 13. PMID 25582849
- [Background] Johns MW. Sleepiness in different situations measured by the Epworth Sleepiness Scale. Sleep. 1994 Dec;17(8):703-10. doi: 10.1093/sleep/17.8.703. PMID 7701181
- [Background] Karkoulias K, Lykouras D, Sampsonas F, Karaivazoglou K, Sargianou M, Drakatos P, Spiropoulos K, Assimakopoulos K. The impact of obstructive sleep apnea syndrome severity on physical performance and mental health. The use of SF-36 questionnaire in sleep apnea. Eur Rev Med Pharmacol Sci. 2013 Feb;17(4):531-6. PMID 23467954
- [Background] Kryger MH, Roth T, Dement WC. Principles and Practice of Sleep Medicine. 5st ed. Elsevier; 2011.
- [Background] Kushida CA, Littner MR, Morgenthaler T, Alessi CA, Bailey D, Coleman J Jr, Friedman L, Hirshkowitz M, Kapen S, Kramer M, Lee-Chiong T, Loube DL, Owens J, Pancer JP, Wise M. Practice parameters for the indications for polysomnography and related procedures: an update for 2005. Sleep. 2005 Apr;28(4):499-521. doi: 10.1093/sleep/28.4.499. PMID 16171294
- [Background] Ieto V, Kayamori F, Montes MI, Hirata RP, Gregorio MG, Alencar AM, Drager LF, Genta PR, Lorenzi-Filho G. Effects of Oropharyngeal Exercises on Snoring: A Randomized Trial. Chest. 2015 Sep;148(3):683-691. doi: 10.1378/chest.14-2953. PMID 25950418
- [Background] Lim YH, Choi J, Kim KR, Shin J, Hwang KG, Ryu S, Cho SH. Sex-specific characteristics of anthropometry in patients with obstructive sleep apnea: neck circumference and waist-hip ratio. Ann Otol Rhinol Laryngol. 2014 Jul;123(7):517-23. doi: 10.1177/0003489414526134. PMID 24668052
- [Background] Logan AG, Perlikowski SM, Mente A, Tisler A, Tkacova R, Niroumand M, Leung RS, Bradley TD. High prevalence of unrecognized sleep apnoea in drug-resistant hypertension. J Hypertens. 2001 Dec;19(12):2271-7. doi: 10.1097/00004872-200112000-00022. PMID 11725173
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- [Background] Martinez D, Gonçalves SC, Fuchs FD. Hipertensão arterial resistente e apneia do sono. Rev Bras Hipertens 2009; 16(3):178-182. Disponível em: <http://departamentos.cardiol.br/dha/revista/16-3/10-hipertensao.pdf>.
- [Background] McNicholas WT. Diagnosis of obstructive sleep apnea in adults. Proc Am Thorac Soc. 2008 Feb 15;5(2):154-60. doi: 10.1513/pats.200708-118MG. PMID 18250207
- [Background] Minayo MC, Hartz ZM, Buss PM. Qualidade de vida e saúde: um debate necessário. Ciência & Saúde Coletiva 2000; 5(1): 7-18. Disponível em: <http://www.scielo.br/scielo.php?script=sci_arttext&pid=S1413-81232000000100002&lng=en&nrm=iso&tlng=pt>
- [Background] Mollayeva T, Thurairajah P, Burton K, Mollayeva S, Shapiro CM, Colantonio A. The Pittsburgh sleep quality index as a screening tool for sleep dysfunction in clinical and non-clinical samples: A systematic review and meta-analysis. Sleep Med Rev. 2016 Feb;25:52-73. doi: 10.1016/j.smrv.2015.01.009. Epub 2015 Feb 17. PMID 26163057
- [Background] Muxfeldt ES, Nogueira Ada R, Salles GF, Bloch KV. Demographic and clinical characteristics of hypertensive patients in the internal medicine outpatient clinic of a university hospital in Rio de Janeiro. Sao Paulo Med J. 2004 May 6;122(3):87-93. doi: 10.1590/s1516-31802004000300003. Epub 2004 Sep 16. PMID 15448805
- [Background] Muxfeldt ES, Margallo VS, Guimaraes GM, Salles GF. Prevalence and associated factors of obstructive sleep apnea in patients with resistant hypertension. Am J Hypertens. 2014 Aug;27(8):1069-78. doi: 10.1093/ajh/hpu023. Epub 2014 Apr 4. PMID 24705438
- [Background] Nadeem R, Molnar J, Madbouly EM, Nida M, Aggarwal S, Sajid H, Naseem J, Loomba R. Serum inflammatory markers in obstructive sleep apnea: a meta-analysis. J Clin Sleep Med. 2013 Oct 15;9(10):1003-12. doi: 10.5664/jcsm.3070. PMID 24127144
- [Background] Netzer NC, Stoohs RA, Netzer CM, Clark K, Strohl KP. Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. Ann Intern Med. 1999 Oct 5;131(7):485-91. doi: 10.7326/0003-4819-131-7-199910050-00002. PMID 10507956
- [Background] NICE - National Institute for Health and Care Excellence.Continuous positive airway pressure for the treatment of sleep apnoea/hypopnoea syndrome. Technology appraisal 139; 2008
- [Background] Nishiyama T, Mizuno T, Kojima M, Suzuki S, Kitajima T, Ando KB, Kuriyama S, Nakayama M. Criterion validity of the Pittsburgh Sleep Quality Index and Epworth Sleepiness Scale for the diagnosis of sleep disorders. Sleep Med. 2014 Apr;15(4):422-9. doi: 10.1016/j.sleep.2013.12.015. Epub 2014 Feb 22. PMID 24657203
- [Background] Nobre MR. [Quality of life]. Arq Bras Cardiol. 1995 Apr;64(4):299-300. No abstract available. Portuguese. PMID 7495385
- [Background] Nuckton TJ, Glidden DV, Browner WS, Claman DM. Physical examination: Mallampati score as an independent predictor of obstructive sleep apnea. Sleep. 2006 Jul;29(7):903-8. doi: 10.1093/sleep/29.7.903. PMID 16895257
- [Background] Oliveira MFR, Souza TGG, Campiotto AR. Contribuição da fonoaudiologia no tratamento de indivíduos roncadores: relato de um caso. In: MarchesanIQ, Zorzi JL, Gomes ICD. Tópicos em fonoaudiologia 1997/1998. São Paulo: Lovise; 1998. p. 489-501.
- [Background] Palombini Lde O. [Pathophysiology of sleep-disordered breathing]. J Bras Pneumol. 2010 Jun;36 Suppl 2:4-9. doi: 10.1590/s1806-37132010001400003. Portuguese. PMID 20944972
- [Background] Parati G, Lombardi C, Hedner J, Bonsignore MR, Grote L, Tkacova R, Levy P, Riha R, Bassetti C, Narkiewicz K, Mancia G, McNicholas WT; European Respiratory Society; EU COST ACTION B26 members. Position paper on the management of patients with obstructive sleep apnea and hypertension: joint recommendations by the European Society of Hypertension, by the European Respiratory Society and by the members of European COST (COoperation in Scientific and Technological research) ACTION B26 on obstructive sleep apnea. J Hypertens. 2012 Apr;30(4):633-46. doi: 10.1097/HJH.0b013e328350e53b. PMID 22406463
- [Background] Pedrosa RP, Drager LF, Gonzaga CC, Sousa MG, de Paula LK, Amaro AC, Amodeo C, Bortolotto LA, Krieger EM, Bradley TD, Lorenzi-Filho G. Obstructive sleep apnea: the most common secondary cause of hypertension associated with resistant hypertension. Hypertension. 2011 Nov;58(5):811-7. doi: 10.1161/HYPERTENSIONAHA.111.179788. Epub 2011 Oct 3. PMID 21968750
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Background] Persell SD. Prevalence of resistant hypertension in the United States, 2003-2008. Hypertension. 2011 Jun;57(6):1076-80. doi: 10.1161/HYPERTENSIONAHA.111.170308. Epub 2011 Apr 18. PMID 21502568
- [Background] Pinto, JA. Ronco e Apneia do Sono. Rio de Janeiro: Revinter; 2010. p. 2;25;40;60.
- [Background] Pitta BDS, Pessoa AF, Sampaio ALL, et al. Terapia miofuncional oral aplicada a dois casos de síndrome da apneia obstrutiva do sono grave. Arq Int Otorrinolaringol; 2007;3:350-4. Disponível em: <http://www.arquivosdeorl.org.br/conteudo/acervo_port.asp?Id=452.
- [Background] Ryan CM, Bradley TD. Pathogenesis of obstructive sleep apnea. J Appl Physiol (1985). 2005 Dec;99(6):2440-50. doi: 10.1152/japplphysiol.00772.2005. PMID 16288102
- [Background] Samsoon GL, Young JR. Difficult tracheal intubation: a retrospective study. Anaesthesia. 1987 May;42(5):487-90. doi: 10.1111/j.1365-2044.1987.tb04039.x. PMID 3592174
- [Background] Somers VK, White DP, Amin R, Abraham WT, Costa F, Culebras A, Daniels S, Floras JS, Hunt CE, Olson LJ, Pickering TG, Russell R, Woo M, Young T. Sleep apnea and cardiovascular disease: an American Heart Association/American College of Cardiology Foundation Scientific Statement from the American Heart Association Council for High Blood Pressure Research Professional Education Committee, Council on Clinical Cardiology, Stroke Council, and Council on Cardiovascular Nursing. J Am Coll Cardiol. 2008 Aug 19;52(8):686-717. doi: 10.1016/j.jacc.2008.05.002. No abstract available. PMID 18702977
- [Background] Tufik S, Santos-Silva R, Taddei JA, Bittencourt LR. Obstructive sleep apnea syndrome in the Sao Paulo Epidemiologic Sleep Study. Sleep Med. 2010 May;11(5):441-6. doi: 10.1016/j.sleep.2009.10.005. Epub 2010 Apr 1. PMID 20362502
- [Background] Zancanella E, Haddad FM, Oliveira LAMP, et al. Apneia Obstrutiva do Sono e Ronco Primário: Diagnóstico. Projeto Diretrizes. Associação Médica Brasileira e Conselho Federal de Medicina; 2012. Disponível em: <http://www.projetodiretrizes.org.br/diretrizes12/apneia_obstrutiva_do_sono_e_ronco_primario_diagnostico.pdf>.